CLINICAL TRIAL: NCT01616225
Title: Adjuvant Growth Hormone in Infertile Women With Prior Poor IVF Response: a Randomized, Controlled, Open-label Study
Brief Title: Growth Hormone in Poor Responders to IVF Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient/slow patient recruitment
Sponsor: Pacific Centre for Reproductive Medicine (Network)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCRM-001
Record Dates: First submitted 2012-04-10; First posted 2012-06-11 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Infertility
Keywords: Infertility; Poor Responder; In Vitro Fertilization; Growth Hormone
MeSH Terms: conditions — Infertility | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Growth Hormone Supplementation (Active Comparator)
  Interventions: Drug: No Saizen Control (Standard IVF Protocol)
- Luteal Growth Hormone Start (Experimental): Growth hormone starting in the luteal phase of the previous menstrual cycle.
  Interventions: Drug: Saizen (Human Growth Hormone)
- Follicular Growth Hormone Start (Experimental): Starting growth hormone during the follicular phase of the prior menstrual cycle.
  Interventions: Drug: Saizen (Human Growth Hormone)

INTERVENTIONS:
Drug: Saizen (Human Growth Hormone) — Subjects will receive the standard protocol treatment, as well as adjuvant GH. One 3.33 mg vial Human Growth Hormone(10 IU Saizen®) will be self-administered daily by subcutaneous injection. GH treatment will start 14 days before FSH start and will continue until the day of the HCG treatment.
  Arms: Luteal Growth Hormone Start
Drug: Saizen (Human Growth Hormone) — Subjects will receive the standard IVF treatment, as well as adjuvant GH as above. One 3.33 mg vial Human Growth Hormone(10 IU Saizen®) will be self-administered daily by subcutaneous injection. GH treatment will start on the same day as the FSH start and will continue until the day of HCG treatment.
  Arms: Follicular Growth Hormone Start
Drug: No Saizen Control (Standard IVF Protocol) — All patients will be administered an oral contraceptive (Marvelon®). FSH treatment (daily subcutaneous injections of 450 IU Gonal-F®; Serono Canada) must begin 4 days after OCP stop, providing both of the following criteria are met. Pituitary downregulation with GnRH antagonist (Cetrotide®, Serono Canada) 0.25mg daily (subcutaneous injection) and LH (Luveris®, Serono Canada) 75 IU daily (subcutaneous injection) will be initiated when one or both of the following criteria are satisfied. Monitoring will continue until a lead follicle reaches ≥18 mm, at which time HCG (Ovidrel®, Serono Canada) 250 mcg will be administered by subcutaneous injection. Oocytes will be retrieved 36 hours after HCG treatment. Luteal support for the endometrium (90 mg progesterone (8% progesterone gel; Crinone® gel), administered intravaginally once daily) will begin one day after oocyte retrieval and will be maintained at least until day 31 of gestation.
  Arms: No Growth Hormone Supplementation

SUMMARY:
This study (the "Adjuvant Growth Hormone Study") is being done to see the effects of adding Growth Hormone (GH) during fertility treatment (also called in vitro fertilization or IVF). Growth Hormone is a protein that your body normally produces. Growth Hormone can act on several different organs, including the ovaries, where eggs are made. From evidence gathered from studies done by fertility doctors over the years, researchers believe that women who have not become pregnant through IVF in the past might have better results if they go on a course of Growth Hormone during the IVF treatment. However, more research needs to be done to confirm whether adding Growth Hormone is beneficial and also to find out the best time to start Growth Hormone treatment during IVF.

We hope that our Adjuvant Growth Hormone study will help answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* Subject with prior poor response(s) to ovarian stimulation for IVF or ICSI. Poor response is defined as a history of producing fewer than four follicles ≥14 mm in diameter during previous COS cycles where FSH or HMG was used from cycle start at a daily dose of ≥450 IU
* Age ≤ 45 years
* Baseline blood labs, measured within previous month, show fasting blood glucose <6.1 mmol/L and TSH ≤ 5.5 mU/L
* Early follicular phase (Day 2 or Day 3) serum FSH, evaluated in the preceding 6 months
* Subject willing and able to give informed consent

Exclusion Criteria:

* Concurrently enrolled in any other clinical trial
* Previous participation in this study
* Using GnRH agonist in COS protocol
* Any prior early follicular phase serum FSH level ≥12 IU/L
* Use of any of the following is contraindicated or inappropriate: GH, Cetrotide®, FSH, LH or hCG
* Used OCP within the prior month
* Pregnant or lactating
* Untreated hydrosalpinx
* Tobacco smoker
* Diabetic or otherwise at risk of gestational diabetes
* BMI > 38 kg/m2
* Poorly controlled thyroid disease
* Known cancer or prior history of malignancies

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Oocyte yield | Following course of treatment (2-3 weeks)
  To assess the effect of adjuvant GH on the number of mature oocytes recovered from women undergoing COS using a GnRH antagonist protocol.

SECONDARY OUTCOMES:
Pregnancy rate | Approximately 2 weeks following completion of treatment.
  To assess the effect of adjuvant GH on: the proportion of subjects reaching embryo transfer; embryo quality; implantation rate; clinical pregnancy rate evaluated 5 weeks after IVF/ICSI (week 7 of gestation); proportion of subjects with clinical pregnancy; mean (SD) crown-rump length 5 weeks after IVF/ICSI (week 7 of gestation); proportion of subjects with a viable fetus(es) at week 12 of gestation; proportion of subjects with live births; duration of FSH stimulation; ampules of FSH consumed; and safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Centre for Reproductive Medicine, Burnaby, British Columbia, Canada